CLINICAL TRIAL: NCT02042417
Title: Comparison of POC-test-equipment With the Standard Method (Laboratory) at ICU-patients
Brief Title: Comparison of POC-test-equipment With the Laboratory
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Hahn, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INRatio_CoaguChek
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: INR-POC-testing

ARMS (1):
- INRatio2 and CoaguChek (Experimental): one measuring per tool, in case of error: one repetiton
  Interventions: Device: INRatio2 and CoaguChek

INTERVENTIONS:
Device: INRatio2 and CoaguChek

SUMMARY:
We compare two POC-tests (INRario2 and CoaguChek) for the INR with the laboratory. Therefore, we take bloodsamples (capillary and venous blood) and put it on the tool. After the measuring, a number is shown = INR.

We develop a Bland-Altman-plot for the correlation between the tool value and the laboratory value to illustrate the applicability in the clinical daily routine.

DETAILED DESCRIPTION:
Including criteria: ICU-patients from 18-99 years

ELIGIBILITY:
Inclusion Criteria:

18-99 years, ICU patients

Exclusion Criteria:

Lupus erythematodes Anti-Phospholipid-Antikörper

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-02; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of POC-test-equipment with the standard method (laboratory) at ICU-patients | 12 months
  outcome measure: Bland Altman plot

CONTACTS AND LOCATIONS:
Locations (1):
- MUVienna, Vienna, Vienna, Austria